CLINICAL TRIAL: NCT02428166
Title: Corneal Changes After Crosslinking in Keratoconus Patients Compared to the Untreated Fellow Eye
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Mike P. Holzer, Ophthalmologist, FEBO, Heidelberg University
Other Study IDs: S-004/2015
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Keratoconus
Keywords: crosslinking; keratoconus; keratometry; pachymetry; pentacam
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this retrospective study is to assess corneal changes (keratometry, pachymetry) and change in visual acuity (VA) in keratoconus patients after unilateral crosslinking treatment compared to the untreated fellow eye. The corneal measurements obtained preoperatively and 2 to 14 months postoperatively using a Pentacam rotating scheimpflug camera are analyzed. Furthermore, pre-existing or actual ocular pathology or/and ocular surgeries as potential factors involved in treatment outcome are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus patients after unilateral crosslinking treatment

Exclusion Criteria:

* Morphological changes of the cornea caused be ocular infection or trauma (e.g. corneal scarring)
* Other pre-existing corneal surgery (e.g. corneal transplantation, implantation of intrastromal corneal ring segments)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Eligible keratoconus patients aged 18-50 years who underwent unilateral crosslinking treatment in our ophthalmology department and completed a postoperative follow-up of 2-14 months
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-02; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Change in maximum keratometry (Kmax) as measured by the Pentacam HR | after completion of data collection based on the measurements preoperatively and 2-14 months postoperative

SECONDARY OUTCOMES:
Change in corneal thickness as measured by the Pentacam HR | retrospective analysis from preoperatively to 2-14 months postoperatively
Change in visual acuity (VA) | retrospective analysis from preoperatively to 2-14 months postoperatively
Evaluation of pre-existing ocular pathology or/and ocular surgery as potential factors involved in treatment outcome | retrospective analysis from preoperatively to 2-14 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Mike P Holzer, MD, FEBO, Principal Investigator — Department of ophthalmology, University of Heidelberg
Locations (1):
- Department of ophthalmology, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany